CLINICAL TRIAL: NCT00465361
Title: Evaluation of Resident Surveillance of Pediatric Patient Developmental Status at the Two Month Preventive Care Visit
Brief Title: Resident Surveillance of Pediatric Patient Developmental Status at the Two Month Preventive Care Visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Sarah Nyp, Medical Physician, Children's Mercy Hospital Kansas City
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 07 02-027E
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Results first posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2011-12

CONDITIONS: Growth & Development; Child Development; Internship and Residency; Education, Medical; Developmental Disabilities
Keywords: Growth and Development; Child Development; Developmental Surveillance; Medical Education; Internship and Residency
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baseline Performance (No Intervention): Observation of baseline performance
- Post-intervention Performance (Experimental): Observation of performance post-intervention
  Interventions: Procedure: performance feedback with an educational module

INTERVENTIONS:
Procedure: performance feedback with an educational module — individual performance feedback with an educational module
  Arms: Post-intervention Performance

SUMMARY:
The purpose of this study is to evaluate the efficacy of individualized performance feedback coupled with an educational module in improving resident performance of the physical and developmental examination component of developmental surveillance of infants at the two month preventive care visit.

DETAILED DESCRIPTION:
Many children in the United States have developmental or behavioral disabilities. The American Academy of Pediatrics recently published a policy statement outlining recommendations for developmental surveillance and screening of infants and young children. One of the Academy's recommendations was for inclusion of developmental surveillance during all preventive care visits. The five components of developmental surveillance include elicitation and attendance to parental concerns, maintenance of the developmental history, observation of the child through physical and developmental examinations, identification of risk and protective factors, and documentation of surveillance findings and process (referral, follow-up, etc.).

As a result of concerns expressed by the public regarding accountability in medical education and health care, the Accreditation Council for Graduate Medical Education and the American Board of Medical Specialties mandated that training programs shift to a competency based assessment system. The focus of this study will be to assess the impact of performance feedback (based upon video recorded observation) coupled with an educational module on resident demonstration of competency in regard to the physical and developmental examinations component of developmental surveillance of infants at the two month preventive care visit.

ELIGIBILITY:
Inclusion Criteria:

* Categorical pediatric residents in their second year of training at Children's Mercy Hospitals and Clinics who are scheduled to see infants for a two month preventive care visit.

Exclusion Criteria:

* Preventive care visits for infants who have parents/guardians who do not speak English fluently
* Preventive care visits for infants who have a previously identified genetic or other medical syndrome or developmental delay

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah S Nyp, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 2007-July 2008 Location: Academic medical center
Pre-assignment Details: Seven participants were enrolled. Four participants did not complete the study due to personal issues.
Groups:
- Intervention: Performance after receiving feedback and educational module
Period: Baseline Assessment
Arm/Group | Intervention
Started | 7
Completed | 3
Not Completed | 4
Not completed — Personal Issues/Scheduling | 4
Period: Post-Intervention Assessment
Arm/Group | Intervention
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Presence of Resident Surveillance Behaviors of Specific Aspects of Developmental Status at the Two Month Preventive Care Visit
Description: Residents were observed to determine whether specific aspects of infant developmental status, as part of developmental surveillance, were assessed during the two-month preventive care visit. The components of developmental surveillance observed were: assessment of the infant's ability to follow past midline, assessment of the infant's ability to lift his/her head off of the table in prone, assessment of the infant's ability to hold an object placed in his/her hand, assessment of the infant's ability to coo, and assessment of the infant's ability to demonstrate a social smile.
Time Frame: Residents were observed during each of the eligible preventive care visits. Each visit was an average of 20 minutes in length. Preventive care visits were observed over a 13 month time period.
Measure: Number; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: May 2007-July 2008
Description: No serious or non-serious adverse events were assessed.
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Long-term effects of intervention are unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes